CLINICAL TRIAL: NCT05068518
Title: The Role of Airway Microbiota on Clinical Phenotypes and Disease Severity in Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin, Chun-Yu, M.D, Chang Gung Memorial Hospital
Other Study IDs: MOST 110-2635-B-182A-006
Record Dates: First submitted 2021-09-28; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
Bronchiectasis is characterized pathologically by permanent bronchial dilatation and airway inflammation. The pathogenesis of the disease and the inflammatory, infective and molecular drivers of disease progression are not fully understood. The concept of "treatable traits" was proposed as biomarker-directed approach, based on the recognition of clinical phenotype and endotypes, help to personalized treatment options. Airway microbiota, including bacteria, NTM and fungus, have important but different inflammatory process in bronchiectasis. Our study will provide a new concept that airway microbiota might involve in the airway and systemic inflammation, mucus hypersecretion, as well as the airway damage, remodeling, and frequent exacerbations in bronchiectasis, thus leading to the deterioration of disease severity.

Bronchiectasis remains a major cause of respiratory morbidity and treatment is generally only partly successful. Our study will give more clues about the mechanisms on the inflammatory pathway and the probably different response among patients with different isolated microbiota from airways.

DETAILED DESCRIPTION:
Bronchiectasis is characterized pathologically by permanent bronchial dilatation and airway inflammation, and clinically by productive cough, hemoptysis and periodic infectious exacerbations. The pathogenesis of the disease and the inflammatory, infective and molecular drivers of disease progression are not fully understood. Current available therapeutic options have shown only a modest impact on disease outcomes in randomized clinical trials. The concept of "treatable traits" was proposed as biomarker-directed approach, based on the recognition of clinical phenotype and endotypes, help to personalized treatment options. Potential treatable traits of airways disease into four broad categories: pulmonary, extra-pulmonary, etiological, and behavior and lifestyle treatable traits. Airway microbiota, including bacteria, NTM and fungus, have important but different inflammatory process in bronchiectasis. Our study will provide a new concept that airway microbiota might involve in the airway and systemic inflammation, mucus hypersecretion, as well as the airway damage, remodeling, and frequent exacerbations in bronchiectasis, thus leading to the deterioration of disease severity.

Bronchiectasis remains a major cause of respiratory morbidity and treatment is generally only partly successful. Our study will give more clues about the mechanisms by which the immunomodulatory medications (macrolides) on the inflammatory pathway and the probably different response among patients with different isolated microbiota from airways. Thus, our results will not only shed light on the airway microbiota inflammatory mechanisms responsible for disease severity, but also provide a new therapeutic direction.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were as follows: bronchiectasis documented on chest HRCT, idiopathic etiology of bronchiectasis, chronic sputum production (daily sputum ≥ 10 ml), absence of other major pulmonary diagnoses, and steady state defined by the absence of change of symptoms noted by the patient over the past 3 weeks

Exclusion Criteria:

* The exclusion criteria were as follows: bronchiectasis with defined etiology (i.e, post-tuberculosis, primary ciliary dyskinesia, allergic bronchopulmonary aspergillosis), common variable immunodeficiency, and use of antibiotics within the last 3 weeks. Patients with hepatic failure, malignancy, or pregnancy were also excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients (age ≥ 20 years old) with bronchiectasis were recruited from the Thoracic Outpatient Clinic of Chang Gung Memorial Hospital in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute exacerbation | one year
  visit ER or hsopitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided